CLINICAL TRIAL: NCT06976541
Title: Utilization Study and Impact Evaluation of the Therapeutic Initiative's Prescribing Portrait and Therapeutics Letter on HbA1c Testing
Brief Title: Utilization Study and Evaluation of Educational Intervention on HbA1c Testing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Ministry of Health, British Columbia (Other Government)
Responsible Party: Principal Investigator, Colin Dormuth, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: H25-01146
Record Dates: First submitted 2025-04-24; First posted 2025-05-16 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: T2DM (Type 2 Diabetes Mellitus); Quality Improvement; Clinical Audit
Keywords: Randomized controlled trial; Type 2 diabetes; HbA1c testing; Quality Improvement; Prescribing Feedback
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The investigators randomized actively practicing family physicians and nurse practitioners into two groups, n=3888 in each group. Investigators then looked at who was registered to access online prescribing Portraits at the time of generating the early Portrait data. Group 1 (n=484) and Group 2 (n=484) for a total of 968 individuals.
  Group 1 received the intervention materials on March 31, 2025, while Group 2 received nothing (control group). Group 2 will receive the intervention materials in 12 months, in March 2026.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Group 1) - Early Portrait + Letter (Experimental): This arm gained access to the prescribing portrait and Therapeutics Letter on March 31, 2025. The materials were uploaded to the Portrait program online portal on this date, and recipients who are registrants to the Portrait program were sent an email notifying them of the new material available.
  Interventions: Behavioral: Portrait + Therapeutics Letter - EARLY
- Arm B (Group 2) - Delayed control (Experimental): This "delayed" control group will get access to the prescribing Portrait and Therapeutics Letter 12 months after Group 1 (March 31, 2026). The materials will be uploaded to the Portrait program online portal on this date, and recipients who are registrants to the Portrait program will be sent an email notifying them of the new material available.
  Interventions: Behavioral: Portrait + Therapeutics Letter - DELAYED
- Arm C (Group 3) - Non-Portrait users (No Intervention): This group will not have access to the Portrait and Therapeutics Letter intervention because they are not registered with the Portrait program (i.e., non Portrait users).

INTERVENTIONS:
Behavioral: Portrait + Therapeutics Letter - EARLY — In the context of audit and feedback interventions, the prescribing Portrait is a document produced by the Therapeutics Initiative that provides personalized prescribing feedback for clinicians in British Columbia. Portraits are used as a practice resource tool for reflection on prescribing or test-ordering patterns. Each Portrait topic provides data of individual prescriber's ordering of HbA1c tests within 90 days of a previous test along with evidence-based benchmarks or targets. Prescribers are also given access to a succinct review of the best available evidence on the topic and recommendations for future action in the Therapeutics Letter, a stand-alone publication that details the evidence for the recommended practice in a brief and practical manner. Therapeutics Letters include a systematic literature review on a clinical topic, and provide references for the data presented in the prescribing Portraits.
  Arms: Arm A (Group 1) - Early Portrait + Letter
Behavioral: Portrait + Therapeutics Letter - DELAYED — In the context of audit and feedback interventions, the prescribing Portrait is a document produced by the Therapeutics Initiative that provides personalized prescribing feedback for clinicians in British Columbia. Portraits are used as a practice resource tool for reflection on prescribing or test-ordering patterns. Each Portrait topic provides data of individual prescriber's ordering of HbA1c tests within 90 days of a previous test along with evidence-based benchmarks or targets. Prescribers are also given access to a succinct review of the best available evidence on the topic and recommendations for future action in the Therapeutics Letter, a stand-alone publication that details the evidence for the recommended practice in a brief and practical manner. Therapeutics Letters include a systematic literature review on a clinical topic, and provide references for the data presented in the prescribing Portraits.
  Arms: Arm B (Group 2) - Delayed control

SUMMARY:
The aim of this randomized trial is to learn if educational materials and personalized prescribing Portraits change the frequency of ordering HbA1c tests by clinicians in British Columbia, Canada.

The main research question: To investigate the overall utilization patterns of HbA1c testing and evaluate the effectiveness of a personalized prescribing Portrait and educational materials to reduce over-utilization of HbA1c tests in diabetes management.

Participants are nurse practitioners and family physicians actively practicing in British Columbia. Participants are registered for the online prescribing Portrait program on the Therapeutics Initiative website where they can access their digital prescribing Portraits. Participants were randomized to receive educational materials on the topic of HbA1c testing either in an Early Group (Group 1 or Arm A) or in a Delayed Group (Group 2 or Arm B). Using administrative health data, the ordering of HbA1c tests by those in the Early Group will be compared with those in the Delayed Group to see if the materials influence the frequency of ordering HbA1c tests. Group 3 (Arm C) will be a control group for Groups 1 and 2 and include participants who receive no intervention.

DETAILED DESCRIPTION:
Diabetes is a major health issue in Canada; about 30% of Canadians are diagnosed with diabetes or prediabetes, with an estimated healthcare system cost of $18.25 billion in 2024.

The glycated Hemoglobin (HbA1c) test is widely used for screening and monitoring diabetes and prediabetes. Canadian guidelines recommend a minimum of 3-month interval for re-testing in diabetes, and 6 months for patients who have reached stable glycemic control. HbA1c test reflects best the blood glucose level in the last 60 to 90 days. Testing too frequently creates unnecessary healthcare costs and burdens for patients and healthcare providers. Testing too infrequently is associated with inadequate glycemic control, and can lead to undiagnosed diabetes and diabetes complications.

Audit and feedback is an approach where individual prescribers receive feedback on their own prescribing or ordering of tests with the aim of improving their prescribing or ordering decisions. The Therapeutics Initiative research group does regular work in this area through the prescribing Portrait program, which aims to improve prescribing by providing audit and feedback and education to prescribers in British Columbia, Canada.

This study is a randomized trial testing the effectiveness of personalized prescribing Portraits and Therapeutics Letters to reduce the over utilization of HbA1c testing for patients with diabetes in the primary care setting in British Columbia. Patients with diabetes will be categorized in 3 groups: 1) diabetes; 2) pre-diabetes; 3) non-diabetic.

7776 active BC clinicians (family physicians and nurse practitioners) were randomly divided into 2 groups (n =3,888 in each group). At the time the Portraits were generated there were 968 people registered for the Portrait program and eligible to access this prescribing Portrait through the secure website (Group 1, n = 484; Group 2, n = 484). A third group of participants who are not registered with the Portrait program and will not have access to the intervention will be compared with Groups 1 and 2 in 2027.

On March 31, 2025 clinicians in Group 1 were notified by email that their prescribing Portraits and Therapeutics Letter were available for viewing in their Portrait accounts. Twelve months later, in March 2026, clinicians in Group 2 will receive this same notification and access to the same materials. The analysis will assess whether the materials led Group 1 clinicians to change how they order HbA1c tests for patients with diabetes.

The analysis will identify:

* Baseline characteristics: Physicians and patients by study group (age, age groups, and sex). Patients with diabetes will be identified with a lookback of 12 months (from January 1, 2022) and will be divided into three categories: 1) diabetes; 2) prediabetes, or 3) non-diabetic.
* Primary outcome: Difference in the change from baseline in the mean number of HbA1c tests per patient. Analysis will use a 2-sample t-test with an α = 0.05 to test whether the difference in the change from baseline is statistically significant.
* Secondary outcome: Difference in the proportion of HbA1c tests ordered within 90 days of another test. The investigators will report relative risk and difference in proportions (with accompanying 95% confidence intervals).

Analysis will be conducted using secondary data from administrative databases from the BC Ministry of Health (under an Information Sharing Agreement). The data are patient level and include anonymized information about demographics, health costs, physician billing codes, prescriptions, outpatient records, and hospitalizations. The data do not include personally identifiable patient information.

ELIGIBILITY:
Inclusion Criteria:

Physicians and nurse practitioners:

* Registered with the College of Physicians and Surgeons of B.C. or BC College of Nurses and Midwives as a nurse practitioner.
* For physicians: defined as a General Practitioner or FP - Emergency Medicine according to the B.C. Ministry of Health's Medical Services Plan (MSP) with a licence status of private practice, temporary licence, salaried, or post graduate.
* Had ≥100 patients with prescriptions filled at a community pharmacy in 2022.

Exclusion Criteria:

* Not registered with the College of Physicians and Surgeons of B.C. or BC College of Nurses and Midwives as a nurse practitioner.
* Physicians who were not classified as a General Practitioner or Family Practice - Emergency Medicine according to the B.C. Ministry of Health's Medical Services Plan (MSP) with a licence status of private practice, temporary licence, salaried, or post graduate.
* Had fewer than 100 patients with prescriptions filled at a community pharmacy in 2023.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 968 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Intention-to-treat analysis | Assessed from 90 days before Jan 1, 2023 to 90 days after Dec 31, 2023 for Group 1. For Group 2, assessed from 90 days prior to Jan 1, 2024 to 90 days after Dec 31, 2024 (12 months + 180 days for both groups).
  The primary outcome is the difference in the change from baseline in the mean number of HbA1c tests ordered per patient.

SECONDARY OUTCOMES:
Intention-to-treat analysis | Assessed from 90 days before Jan 1, 2023 to 90 days after Dec 31, 2023 for Group 1. For Group 2, assessed from 90 days prior to Jan 1, 2024 to 90 days after Dec 31, 2024 (12 months + 180 days for both groups).
  The secondary outcome is the difference in the proportion of HbA1c tests ordered within 90 days of another test.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Dormuth, ScD, Principal Investigator — University of British Columbia
Locations (1):
- Therapeutics Initiative - Dept of Anesthesiology, Pharmacology & Therapeutics, Faculty of Medicine, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
The data access agreement for the Therapeutics Initiative does not permit sharing of IPD.

REFERENCES:
- See also: Therapeutics Initiative website which describes the Portrait program in more detail. — https://www.ti.ubc.ca/portrait/